CLINICAL TRIAL: NCT06281795
Title: Neuromodulation of the Autonomic Nervous System in Athletes (NANSA Trial)
Brief Title: Neuromodulation of the Autonomic Nervous System in Athletes
Acronym: NANSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bakulev Scientific Center of Cardiovascular Surgery (Other Government)
Collaborators: Foundation for the Support of Physical Culture and Sports BECOME A CHAMPION (Unknown); Autonomous Non-Profit organization of additional education sports school BECOME A CHAMPION (Unknown)
Responsible Party: Principal Investigator, Vladimir A Shvartz, MD, MD, DM, Professor, Bakulev Scientific Center of Cardiovascular Surgery
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1.24.
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Efficacy, Self; Fatigue; Muscle, Heart; Fatigue, Mental; Fatigue; Combat
Keywords: auricular stimulation; auricular vagus nerve stimulation; transcutaneous vagus nerve stimulation (tVNS); vagus nerve stimulation (VNS); heart rate; heart rate variability; power of high-frequency oscillations (HF); power of low-frequency oscillations (LF); LF/HF; index centralization (IC); index of vegetative balance (IVB); athletes; sport; maximum oxygen consumption (VO2max); treadmill speed; anaerobic threshold of metabolism.; aerobic metabolism threshold of metabolism
MeSH Terms: conditions — Fatigue; Mental Fatigue; Combat Disorders

STUDY DESIGN:
Intervention Model Description: 1:1 randomization of active stimulation vs. sham stimulation
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tVNS (Active Comparator): Active stimulation will be carried out using the tVNS device with an ear clip attached to the tragus of the left ear at a frequency of 20 Hz, 200 μs at a current slightly below the discomfort threshold. The device's operating mode is active therapeutic.
  Interventions: Device: tVNS
- Sham tVNS (Sham Comparator): Fictitious stimulation will be carried out using the tVNS device with an ear clip attached to the tragus of the left ear at a frequency of 20 Hz, 200 μs at a current slightly below the discomfort threshold. The device's operating mode is research mode.
  Interventions: Device: tVNS

INTERVENTIONS:
Device: tVNS — tVNS will be performed daily after workouts for 60 minutes over a period of 8 weeks.

SUMMARY:
There are few studies in the literature that have evaluated the effects of using percutaneous stimulation of the auricular branch of the vagus nerve for sports purposes (to accelerate recovery after physical exertion). It has been demonstrated that tVNS in athletes improved the rate of heart rate recovery, reduced lactic acid levels in blood plasma, reduced pain, reduced overtraining syndrome and fatigue levels.

DETAILED DESCRIPTION:
Several studies have shown that transcutaneous vagus nerve stimulation (tVNS) potentially exhibits therapeutic effects similar to its invasive counterpart. tVNS is performed using surface electrodes and low-frequency electrical currents, targeting specific locations, most commonly the auricular branch of the vagus nerve or its cervical branch.

Stimulation of the auricular branch of the vagus nerve activates vagal sensory fibers, simulating sensory input to the brainstem and forming what is known as the auriculo-vagal afferent pathway. Since these fibers project directly to the nucleus of the solitary tract (also known as the solitary tract nucleus), which in turn has direct or indirect projections to nuclei that provide noradrenergic, endorphinergic, and serotonergic fibers in various parts of the brain, regulating systemic parameters of cardiovascular, respiratory, and immune functions, it can be expected that the body's response to stimulation of the auricular branch of the vagus nerve will be systemic.

With the onset of physical exercise, sympathetic activity in the body increases and reaches a plateau value after a certain period of maximum activity. After the end of physical exercise, suppressed parasympathetic activity begins to intensify, and the sympathetic system gradually returns to a resting state. After training, parasympathetic system activation continues for up to 48 hours. In certain types of training, when the frequency of anaerobic respiration increases during physical exertion, a decrease in parasympathetic reactivation may be observed.

In the literature, there are individual studies that have evaluated the effects of transcutaneous stimulation of the auricular branch of the vagus nerve for sports purposes (to accelerate recovery processes after physical exertion). It has been demonstrated that tVNS in athletes improves heart rate recovery, reduces lactate levels in plasma, reduces pain sensations, decreases overtraining syndrome, and reduces fatigue levels.

The aim of this study is to: evaluate the influence of low-frequency electrical stimulation of the auricular branch of the vagus nerve on the functional reserve of the cardiovascular and respiratory systems in athletes during the post-training period, after high-intensity workouts.

ELIGIBILITY:
Inclusion Criteria:

* Professional athletes over the age of 15 and under the age of 35;
* Cyclic sports (swimming, modern pentathlon, athletics, triathlon);
* Difficult coordination sports (dance sports, rhythmic gymnastics);
* Sports category: no lower than candidate for master of sports;
* Voluntary informed consent.

Exclusion Criteria:

* Atypical and unrelated to physical exertion changes on the ECG (T wave inversion, st-segment depression, pathological Q waves, signs of left atrial enlargement, signs of right ventricular hypertrophy, ventricular pre-excitation, complete right or left bundle branch block, prolonged or shortened Q-T interval, Brugada-like early repolarization);
* Heart rhythm and conduction disorders (frequent ventricular and supraventricular extrasystoles, first-degree atrioventricular block (P-Q > 0.21 s, not shortened during hyperventilation or physical exertion), second or third degree);
* Expressed sinus bradycardia with resting heart rate < 40 bpm;
* Taking glucocorticosteroids in the last 1 month;
* Taking any antiarrhythmic drugs, including beta-blockers.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Dynamics of maximum oxygen consumption (VO2max). | The level of VO2max is estimated at the beginning of the study (initially) and at the end of the study (after 8 weeks) in the active and fictitious stimulation groups.
  During a cardiorespiratory exercise test, the level of VO2max (ml/min/kg) is assessed.
The dynamics of the treadmill speed at the level of the anaerobic threshold of metabolism. | Treadmill speed is estimated at the beginning of the study (initially) and at the end of the study (after 8 weeks) in the active and dummy stimulation groups.
  During the cardiorespiratory exercise test, the treadmill speed (km/h) is estimated at the level of the anaerobic metabolic threshold.

SECONDARY OUTCOMES:
Dynamics of the treadmill speed at the level of the aerobic metabolism threshold of metabolism. | Treadmill speed is estimated at the beginning of the study (initially) and at the end of the study (after 8 weeks) in the active and dummy stimulation groups.
  During the cardiorespiratory exercise test, the treadmill speed (km/h) is estimated at the level of the aerobic metabolic threshold.
The dynamics of the heart rate (HR) at the level of the anaerobic threshold of metabolism. | HR is estimated at the beginning of the study (initially) and at the end of the study (after 8 weeks) in the active and dummy stimulation groups.
  During the cardiorespiratory exercise test, the HR is estimated at the level of the anaerobic metabolic threshold.
The dynamics of the heart rate (HR) at the level of the aerobic threshold of metabolism. | HR is estimated at the beginning of the study (initially) and at the end of the study (after 8 weeks) in the active and dummy stimulation groups.
  During the cardiorespiratory exercise test, the HR is estimated at the level of the aerobic metabolic threshold.
The dynamics of RMSSD. | This parameter is evaluated at the beginning of the study (initially) and at the end of the study (after 8 weeks) in the groups of active and fictitious stimulation.
  During the time analysis of heart rate variability, the RMSSD parameter is estimated.
HF dynamics | This parameter is evaluated at the beginning of the study (initially) and at the end of the study (after 8 weeks) in the groups of active and fictitious stimulation.
  During the spectral analysis of heart rate variability, the HF (high frequency) parameter is estimated.
Dynamics of the LF/HF ratio. | This LF/HF ratio is evaluated at the beginning of the study (initially) and at the end of the study (after 8 weeks) in the active and fictitious stimulation groups.
  The LF/HF ratio is estimated during the spectral analysis of heart rate variability.

CONTACTS AND LOCATIONS:
Overall Officials: Vasiliy Danilov, Study Chair — Autonomous Non-Profit organization of additional education sports school BECOME A CHAMPION
Locations (1):
- Autonomous Non-Profit organization of additional education sports school BECOME A CHAMPION, Krasnodar, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The effect of transcutaneous auricular vagus nerve stimulation on cycling ergometry and recovery in healthy young individuals — https://pubmed.ncbi.nlm.nih.gov/37974551/